CLINICAL TRIAL: NCT07139028
Title: Effects of Tibialis Anterior Resistance Training With Ladder Drills on Agility, Power and Speed in Basketball Athletes
Brief Title: Effects of Tibialis Anterior Resistance Training With Ladder Drills in Basketball Athletes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0436
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Sports Physical Therapy
Keywords: Ladder; Power; Resistance training; Tibialis muscle; Speed

STUDY DESIGN:
Intervention Model Description: Randomized Control Design
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and assessor are blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tibialis anterior resistance training and ladder drills (Experimental): Group A (Experimental):
  19 participants will be in experimental group A, they will perform tibialis anterior resistance training exercises with ladder drills (3 times/ week for 6 weeks) along with traditional training
  Interventions: Other: Tibialis Anterior resistance training and ladder drills
- Traditional training (Experimental): Group B (Control):
  19 participants will be in control group B,they will perform only traditional training (guided by coach)
  Interventions: Other: Traditional training

INTERVENTIONS:
Other: Tibialis Anterior resistance training and ladder drills — 19 participants will be in experimental group A, they will perform tibialis anterior resistance training exercises with ladder drills (3 times/ week for 6 weeks) along with traditional training
  Arms: Tibialis anterior resistance training and ladder drills
Other: Traditional training — 19 participants will be in control group B,they will perform only traditional training (guided by coach)
  Arms: Traditional training

SUMMARY:
The effects of tibialis anterior resistance training with ladder drills in basketball athletes.

DETAILED DESCRIPTION:
The effects of tibialis anterior resistance training with ladder drills on agility, power and speed in basketball athletes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 30 years
* Minimum 2 years of basketball experience
* Able to perform agility drills
* No significant lower extremity injury in past 6 months

Exclusion Criteria:

* Current or past ankle or knee instability or pain
* Past surgical history (involving knee or ankle)
* Past medical history (heart condition, neurological condition)
* Players with recent history of concussion injury (past 3 months)
* Taking any medication (muscle relaxant or anti-inflammatory drugs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Illinois agility test: ( for agility) | 6 weeks
  The Illinois agility test (IAT) is a comprehensive agility test used to assess an athlete's agility and quickness. This test will include the following components, start and finish lines, zigzag running between cones, shuttle-run between cones, figure 8 runs around cones and 10-yard dash. This test is typically performed using stopwatch and total time of course to complete is recorded. The faster the time the better the agility score, the validity of illinois test is 0.95 and reliability is 0.95.
20-meter sprint test: (for speed) | 6 weeks
  20-meter sprint test is used to assess speed in athletes over a short distance. The total distance which is 20-meter covered in amount of time is measured using a stopwatch and the time recorded determines the speed of an athlete. The validity of this test is 0.80 and reliability of 0.95.
Vertical jump test: (for power) | 6 weeks
  A vertical jump test is used to assess the muscular power of an athlete. The athlete is asked to stand with feet shoulder width apart, arms at sides, a point is put at the maximum height of athlete. Then he/she is asked to jump straight from the ground, extending arms and legs. The maximum height reached is recorded from starting point to ending point. The readings should be taken at least 3 times for accuracy. Height measured is typically recorded in centimeters (cm)/inches(inch). The validity of this test is 0.90 and reliability of 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: Meryam Mujahid, DPT, Principal Investigator — Riphah International University
Locations (1):
- YMCA basketball club, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behm DG, Granacher U, Warneke K, Aragao-Santos JC, Da Silva-Grigoletto ME, Konrad A. Minimalist Training: Is Lower Dosage or Intensity Resistance Training Effective to Improve Physical Fitness? A Narrative Review. Sports Med. 2024 Feb;54(2):289-302. doi: 10.1007/s40279-023-01949-3. Epub 2023 Nov 4. PMID 37924459
- [Background] Saeterbakken AH, Stien N, Pedersen H, Langer K, Scott S, Michailov ML, Gronhaug G, Balas J, Solstad TEJ, Andersen V. The Connection Between Resistance Training, Climbing Performance, and Injury Prevention. Sports Med Open. 2024 Jan 19;10(1):10. doi: 10.1186/s40798-024-00677-w. PMID 38240903
- [Background] Cao S, Liu J, Wang Z, Geok SK. The effects of functional training on physical fitness and skill-related performance among basketball players: a systematic review. Front Physiol. 2024 May 9;15:1391394. doi: 10.3389/fphys.2024.1391394. eCollection 2024. PMID 38784117
- [Background] Swinton PA, Schoenfeld BJ, Murphy A. Dose-Response Modelling of Resistance Exercise Across Outcome Domains in Strength and Conditioning: A Meta-analysis. Sports Med. 2024 Jun;54(6):1579-1594. doi: 10.1007/s40279-024-02006-3. Epub 2024 Apr 23. PMID 38652410
- [Background] Parlakidis K, Kontopoulos LA, Mandalidis D, Paraskevopoulos E, Papandreou M, Kapreli E, Christakou A. The Effectiveness of External Verbal Feedback on Balance in Athletes with Chronic Ankle Instability. J Funct Morphol Kinesiol. 2024 Mar 21;9(1):56. doi: 10.3390/jfmk9010056. PMID 38535436
- [Background] Markov A, Hauser L, Chaabene H. Effects of Concurrent Strength and Endurance Training on Measures of Physical Fitness in Healthy Middle-Aged and Older Adults: A Systematic Review with Meta-Analysis. Sports Med. 2023 Feb;53(2):437-455. doi: 10.1007/s40279-022-01764-2. Epub 2022 Oct 12. PMID 36222981
- [Background] Hameed I, Farooq N, Haq A, Aimen I, Shanley J. Role of strengthening exercises in management and prevention of overuse sports injuries of lower extremity: a systematic review. J Sports Med Phys Fitness. 2024 Aug;64(8):807-815. doi: 10.23736/S0022-4707.23.15470-3. Epub 2024 Mar 12. PMID 38470015
- [Background] Pardos-Mainer E, Lozano D, Torrontegui-Duarte M, Carton-Llorente A, Roso-Moliner A. Effects of Strength vs. Plyometric Training Programs on Vertical Jumping, Linear Sprint and Change of Direction Speed Performance in Female Soccer Players: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jan 6;18(2):401. doi: 10.3390/ijerph18020401. PMID 33419178
- [Background] Palermi S, Vittadini F, Vecchiato M, Corsini A, Demeco A, Massa B, Pedret C, Dorigo A, Gallo M, Pasta G, Nanni G, Vascellari A, Marchini A, Lempainen L, Sirico F. Managing Lower Limb Muscle Reinjuries in Athletes: From Risk Factors to Return-to-Play Strategies. J Funct Morphol Kinesiol. 2023 Nov 6;8(4):155. doi: 10.3390/jfmk8040155. PMID 37987491
- [Background] Carvalho L, Junior RM, Barreira J, Schoenfeld BJ, Orazem J, Barroso R. Muscle hypertrophy and strength gains after resistance training with different volume-matched loads: a systematic review and meta-analysis. Appl Physiol Nutr Metab. 2022 Apr;47(4):357-368. doi: 10.1139/apnm-2021-0515. Epub 2022 Jan 11. PMID 35015560